CLINICAL TRIAL: NCT05445700
Title: The Effects of Frailty on Opioid Consumption After Total Knee Arthroplasty
Brief Title: The Effects of Frailty on Opioid Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet SARGIN, Associate professor, Selcuk University
Allocation: Non-Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-1
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Frailty; Opioid Use; Knee Arthropathy
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Groups will be determined according to frailty status.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-frail (Active Comparator): FRAIL scale= 0
  Interventions: Device: Patient-controlled analgesia pump (PCA)
- Pre_frail (Active Comparator): FRAIL scale= 1-2
  Interventions: Device: Patient-controlled analgesia pump (PCA)
- Frail (Active Comparator): FRAIL scale >2
  Interventions: Device: Patient-controlled analgesia pump (PCA)

INTERVENTIONS:
Device: Patient-controlled analgesia pump (PCA) — Each patient will receive a PCA pump with intravenous (i.v.) morphine.

SUMMARY:
The FRAIL scale will be applied to patients at the preoperative visit. According to the FRAIL Scale, patients will be divided into 3 groups as Non-frail (Group I), pre-frail (Group II) and frail (Group III). After routine preoperative preparation and monitoring, patients will be given spinal anesthesia. Demographic data and intraoperative data of the patients will be recorded. Patients will be transferred to the post-operational post-operative care unit (PACU) and patient-controlled analgesia (PCA) will be applied to each patient with a standard protocol. In the postoperative period, the need for analgesics will be recorded for 24 hours, and if additional analgesics are needed, they will be recorded. Pain scores of the patients will be evaluated for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo unilateral, primary total knee arthroplasty
* Patients who will be operated with spinal anesthesia

Exclusion Criteria:

* Patients with ASA IV and above physical status
* Uncooperative patients
* Patients who do not speak Turkish
* Patients on routine opioid use

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Postoperative 24th hour
  Total opioid consumption (24 hours)

SECONDARY OUTCOMES:
Visual analog pain scores (VAS) | 6,12 and 24 hours
  VAS scores will evaluate at rest and during 45° active knee flexion
Nausea and vomiting questionnaire | Postoperative for 24 hours
  Postoperative nausea and vomiting will be evaluated by asking the patient whether she/he has had nausea and vomiting for 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Medical Faculty Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No